CLINICAL TRIAL: NCT02189642
Title: Evaluation of Perioperative Outcomes in Children: Creation of the Boston Children's Hospital Perioperative Outcomes Registry
Brief Title: Boston Children's Hospital Post Anesthesia Care Unit Outcomes Study
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph P. Cravero, Department of Anesthesiology, Senior Associate, Boston Children's Hospital
Other Study IDs: IRB-P00008050
Record Dates: First submitted 2014-07-11; First posted 2014-07-14 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Genito-Urinary/Urology Surgical Procedure Types: Pediatric patients undergoing circumcision, orchidopexy, hypospadias repair, hernia repair, cystoscopy, pyeloplasty, and ureteral reimplants or ureteral stents.
- Otolaryngology Surgical Procedure Types: Pediatric patients undergoing tonsil and/or adenoid removal, tympanostomy, tympanoplasty, and mastoidectomy.
- Orthopaedics Surgical Procedure Types: Patients undergoing hip and knee arthroscopies, hardware removal, and tendon lengthening.
- Plastic Surgery Surgical Procedure Type: Pediatric patients undergoing alveolar cleft repair.

SUMMARY:
The purpose of this study is to evaluate the quality of outcomes in the Post Anesthesia Care Unit (PACU) at BCH and to identify preoperative demographic and behavioral data as well as intraoperative and anesthetic predictors of adverse PACU outcomes. The investigators hypothesize quality of PACU outcomes will correlate with preoperative demographic and behavioral characteristics as well as intraoperative and anesthetic procedures/techniques. This study will help the investigators improve post anesthetic care quality and create a higher level of satisfaction for patients, family, and health care providers.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for surgery at Boston Children's Hospital ages 6 months to 30 years undergoing the following qualifying surgeries:

Genito-Urinary/Urology Department:

* Circumcision, Orchidopexy, Hypospadias Repair, Hernia Repair, Cystoscopy, Pyeloplasty, and Ureteral Reimplants or Ureteral Stents.

Otolaryngology Department:

* Tonsil and/or Adenoid Removal, Tympanostomy, Tympanoplasty, and Mastoidectomy.

Orthopaedics Department:

* Hip and Knee Arthroscopies, Hardware Removal, and Tendon Lengthening.
* Plastic Surgery Department: Alveolar Cleft Repair.

Exclusion Criteria:

* English as a second language.
* < 6 months, > 21 or 30 (hip patients only).
* Resident of a residential facility or ward of state.
* Guardianship status unclear.
* Not headed to the PACU post-operatively.
* Day of: Projected to arrive in PACU after 3 PM.
* Duration of surgery well beyond ordinary for procedure type.
* Exceptionally complex medical history.

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators will enroll all patients ages 6 months to 30 years undergoing the following qualifying surgeries:
  • Genito-Urinary/Urology Department
  Circumcision, Orchidopexy, Hypospadias Repair, Hernia Repair, Cystoscopy, Pyeloplasty, and Ureteral Reimplants or Ureteral Stents
  • Otolaryngology Department
  Tonsil and/or Adenoid Removal, Tympanostomy, Tympanoplasty, and Mastoidectomy
  • Orthopaedics Department
  Hip and Knee Arthroscopies, Hardware Removal, and Tendon Lengthening
  • Plastic Surgery Department
  Alveolar Cleft Repair
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2013-07-13; Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Significant Pain in PACU | On day of surgery.
  Incidence of significant pain defined by pain behavior information from the Faces-Legs-Activity-Cry-Consolability (FLACC) scale, Wong-Baker Faces scale, visual analog scale/numerical scale or adapted numerical rating scale - equal to or more than 5 on a scale from 0 to 10 at any time during the PACU stay.
Incidence of Agitation in PACU | On day of surgery.
  Incidence of agitation using emergence agitation categorization with Pediatric Agitation Emergence Delirium (PAED) scale equal to or more than 10 on this scale for more than 30 seconds during the recovery period.
Incidence of Post-Operative Nausea or Vomiting | On day of surgery.
  Post-operative vomiting (POV) will be measured by episodes of vomiting or retching in PACU. This will be a binary outcome - either vomiting/retching occurred or it did not.

SECONDARY OUTCOMES:
Satisfaction of Patients and Families with Post-Operative Care | At two days and two weeks after surgery.
  Satisfaction of patients and families with perioperative care, as determined from a three-question satisfaction survey allowing participating families to rate their recovery experience, global surgical experience, and need for further care at another healthcare facility.
Post-Hospitalization Behavior Changes | At two days and two weeks after surgery.
  Post-hospitalization behaviors changes defined by development of 4 or more behavior changes on the Post Hospitalization Behavior Questionnaire (PHBQ) or development of increased stress levels on the Child PTSD Symptom Scale (CPSS).

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States